CLINICAL TRIAL: NCT03949335
Title: Clinical Investigation of the Safety and Effectiveness of an Investigational Model of the TECNIS® Intraocular Lens
Acronym: BRAVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUR-CAT-652-2001
Record Dates: First submitted 2019-05-01; First posted 2019-05-14 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the surgeon and the operative staff will know which lens type is implanted and will be unmasked throughout the study. There may also be site coordinators and other site study staff, such as those performing slit-lamp exams, who will be unmasked. Unmasked study staff and study subjects will be instructed not to disclose the lens type the subject received or to talk about the lens to any subjects or masked evaluators.
  The subjects and the study technicians performing the postoperative vision tests are to be masked through study completion. To maintain subject/technician-masking through the 6-month study exams, a masking plan will be tailored for each site to detail how lens assignment information will be concealed from masked technicians.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational (Experimental): Bilateral implantation with investigational IOL Model ZFR00V
  Interventions: Device: IOL Model ZFR00V
- Control (Active Comparator): Bilateral implantation with control IOL Model ZCB00
  Interventions: Device: IOL Model ZCB00

INTERVENTIONS:
Device: IOL Model ZFR00V — Bilateral implantation with Investigational IOL Model ZFR00V
  Arms: Investigational
Device: IOL Model ZCB00 — Bilateral Implantation with control IOL Model ZCB00
  Arms: Control

SUMMARY:
This study will be a prospective, multicenter, bilateral, comparative, three-way masked (Sponsor, subject and evaluator), randomized clinical investigation conducted at up to 15 sites. Up to 300 subjects will be enrolled to achieve approximately 270 bilaterally implanted subjects, resulting in approximately 244 evaluable subjects (122 per lens group) at 6 months. After informed consent is obtained and confirmation that all eligibility criteria are met, the eye(s) may be treated according to randomization.

After signing the informed consent form, subjects meeting all eligibility criteria will be randomized in a masked fashion to a treatment group: either the investigational IOL Model ZFR00V or the control IOL Model ZCB00. Prior to randomization, the investigator will choose which eye to operate on first for each subject at his/her discretion based on his/her standard clinical practice (e.g., the eye with the worse cataract, poorer best corrected distance vision and/or more severe optical/visual complaints). All subjects are intended to have bilateral cataract surgery with the second eye surgery occurring after the 1-week postoperative exam for the first eye, but no more than 30 days after the first eye surgery. All subjects will be examined through 6 months postoperatively according to the visit schedule

ELIGIBILITY:
Inclusion Criteria:

* be at least 22 years old
* have cataracts in both eyes
* sign the written informed consent
* be willing and able to comply with examination procedures
* understand, read and write English to complete informed consent and questionnaires
* be available for study follow-up visits

Exclusion Criteria:

* currently participating in any other clinical study or have participated in a clinical study during the last 60 days
* have a certain disease/illness such as poorly-controlled diabetes
* have certain ocular conditions such as uncontrolled glaucoma
* Is taking medication that may affect vision
* Subject is pregnant, plan to become pregnant during the study, or is breastfeeding

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (15):
- United States (15):
  - Empire Eye & Laser Center, Bakersfield, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Katzen Eye Care & Laser Center, West Palm Beach, Florida
  - Jones Eye Clinic, Sioux City, Iowa
  - Chesapeake Eye Care & Laser Center, Annapolis, Maryland
  - Cincinnati Eye Institute, Blue Ash, Ohio
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Carolina EyeCare Physicians, Mt. Pleasant, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Berkeley Eye Institute, Houston, Texas
  - Texas Eye and Laser Center, Hurst, Texas
  - Lehmann Eye Center, Nacogdoches, Texas
  - Focal Point Vision, San Antonio, Texas
  - Clarus Eye Centre, Lacey, Washington

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu/

REFERENCES:
- [Derived] Chang DH, Hu JG, Lehmann RP, Thompson VM, Tsai LH, Thomas EK. Clinical performance of a hybrid presbyopia-correcting intraocular lens in patients undergoing cataract surgery in a multicenter trial. J Cataract Refract Surg. 2023 Aug 1;49(8):840-847. doi: 10.1097/j.jcrs.0000000000001205. PMID 37097283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 272 subjects were bilaterally implanted with either the study or control lens. 135 subjects were bilaterally implanted with the study lens and 137 subjects were bilaterally implanted with the control lens. All 272 subjects were bilaterally implanted with the same IOL model in both eyes.
Groups:
- ZFR00V: Study Lens
- ZCB00: Control Lens
Period: Overall Study
Arm/Group | ZFR00V | ZCB00
Started | 135 | 137
Completed | 132 | 131
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZFR00V | ZCB00 | Total
Number analyzed (Participants) | 135 | 137 | 272
Age, Customized [Number; unit: Participants]
  <60 | 17 | 17 | 34
  60 to 69 | 50 | 57 | 107
  70 to 79 | 62 | 56 | 118
  > or = 80 | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 90 | 184
  Male | 41 | 47 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 127 | 130 | 257
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (including Indian) | 3 | 1 | 4
  Black | 15 | 19 | 34
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  Caucasian | 114 | 116 | 230
  Other Race | 2 | 1 | 3
  Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distance-Corrected Near Visual Acuity (DCNVA) at 40 cm
Description: mean photopic monocular Distance Corrected Near Visual Acuity results at 40 cm for ZFR00 and control first eyes in the safety population at 6 months
Time Frame: 6 months (postoperative)
Population: The safety (SP) population for monocular Distance-Corrected Near Visual Acuity include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
LogMAR | 0.104 (0.138) | 0.522 (0.193)
Statistical Analysis 1: Comparison: ZFR00V vs ZCB00; Test type: Superiority; p < 0.0001, t-test, 1 sided

2. Secondary Outcome: Monocular Distance-Corrected Intermediate Visual Acuity at 66 cm
Description: mean photopic monocular Distance-Corrected Intermediate Visual Acuity results at 6 months for ZFR00 and control first eyes in the safety population
Time Frame: 6 months (postoperative)
Population: The safety (SP) population for monocular Distance-Corrected Intermediate Visual Acuity include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
LogMAR | 0.060 (0.115) | 0.335 (0.155)
Statistical Analysis 1: Comparison: ZFR00V vs ZCB00; Test type: Superiority; p < 0.0001, t-test, 1 sided

3. Secondary Outcome: Monocular Distance-Corrected Near Visual Acuity at 33 cm
Description: mean photopic monocular Distance-Corrected Near Visual Acuity results at 33 cm for ZFR00 and control first eyes in the safety population at 6 months
Time Frame: 6 months postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
LogMAR | 0.154 (0.151) | 0.608 (0.187)
Statistical Analysis 1: Comparison: ZFR00V vs ZCB00; Test type: Superiority; p < 0.0001, t-test, 1 sided

4. Secondary Outcome: Monocular Photopic Best-Corrected Distance Visual Acuity
Description: mean monocular Best-Corrected Distance Visual Acuity results at 6 months for ZFR00 and control first eyes in the safety population.
Time Frame: 6 months postoperative
Population: The safety (SP) population for monocular Best-Corrected Distance Visual Acuity include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
LogMAR | -0.014 (0.087) | -0.045 (0.089)
Statistical Analysis 1: Comparison: ZFR00V vs ZCB00; Test type: Non-Inferiority — Noninferiority margin equals -0.1; Success criteria was evaluated using lower confidence interval. No P-Value was calculated; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.053 to -0.010]

5. Secondary Outcome: Monocular Distance-Corrected Defocus Curve
Description: Mean monocular (first eye) distance-corrected defocus curve for each lens group at 6 months in the safety population
Time Frame: 6 months postoperative
Population: The safety (SP) population for monocular Distance-Corrected Defocus Curve include all first eyes implanted with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Mean (Full Range); unit: diopter
Units Other Than Participants: Eyes
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
diopter | -3.3 [-3.6 to -3.0] | -0.9 [-1.1 to -0.7]

6. Secondary Outcome: Spectacle Wear
Description: Spectacle wear is determined via the PRO questionnaire instrument and defined as wearing glasses or contacts "none of the time" in all 4 conditions (distance vision, intermediate vision, near vision and overall vision) at 6 months postoperative.
Time Frame: 6 months postoperative
Population: The safety (SP) population for spectacle independence include all subjects implanted bilaterally with either a test or control IOL with data available at 6 months postoperative (i.e., no data imputation)
Measure: Count of Participants; unit: Participants
Arm/Group | ZFR00V | ZCB00
Number analyzed (Participants) | 131 | 131
Participants
  None of the time | 115 | 4
  A little/Some/Most/All of the time | 16 | 127
  Not reported | 0 | 0
Statistical Analysis 1: Comparison: ZFR00V vs ZCB00; Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events (AEs) were planned to be reported for each eye separately and AEs not related to eyes were counted and represented in both the eyes.
  The total number of participants affected by SAE is total number of unique eyes. If an eye has multiple SAEs, the number of affected participant is one (1) but list multiple number of SAEs.
  Only other (not including serious) adverse events that exceed the frequency threshold of 5% are reported.
Groups:
- ZFR00V First Eye; ZFR00V Second Eye: Study Lens
- ZCB00 First Eye; ZCB00 Second Eye: Control Lens
Arm/Group | ZFR00V First Eye | ZCB00 First Eye | ZFR00V Second Eye | ZCB00 Second Eye
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/137 | 0/135 | 0/137
Serious Adverse Events (participants affected / at risk) | 6/135 | 2/137 | 8/135 | 3/137
Other Adverse Events (participants affected / at risk) | 10/135 | 0/137 | 0/135 | 0/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZFR00V First Eye (N=135) | ZCB00 First Eye (N=137) | ZFR00V Second Eye (N=135) | ZCB00 Second Eye (N=137)
Cystoid Macular Edema (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Undesirable Optical Phenomena (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment/tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular Hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Simplex Virus Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic Anterior Segment Syndrome (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal Ulcers (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopyon (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retained lens material resulting in secondary surgical intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Due to high blood pressure and high blood sugar
Fractured right fibula and dislocated ankle requiring surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Exacerbation of congestive heart failure and atrial fibrillation
Abdominal Hernia requiring surgical repair (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Due to pneumonia due to influenza
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZFR00V First Eye (N=135) | ZCB00 First Eye (N=137) | ZFR00V Second Eye (N=135) | ZCB00 Second Eye (N=137)
Undesirable Optical Phenomena (Product Issues) | 10 (10) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03949335/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03949335/SAP_001.pdf